CLINICAL TRIAL: NCT04491071
Title: Stress Induced by the COVID-19 Pandemic and Nonconfinement: Study of Anxiety Factors and Potential Effects on Immunity.
Acronym: SCEI
Status: Terminated | Type: Observational
Why Stopped: The study was stopped due to lack of inclusions
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH129; IRBN972020/CHUSTE (Other: Comité d'éthique)
Record Dates: First submitted 2020-07-27; First posted 2020-07-29 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Stress Disorder
Keywords: COVID-19; Stress; Effects on Immunity; Anxiety
MeSH Terms: conditions — Stress Disorders, Traumatic; COVID-19; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Volunteers: volunteers over 18 years of age
  Interventions: Diagnostic Test: Generalized Anxiety Disorder-7 (GAD 7); Diagnostic Test: Background questionnaire; Diagnostic Test: Impact of COVID-19 questionnaire; Diagnostic Test: Confinement and Communication During the COVID-19 Pandemic; Diagnostic Test: Mental Health questionnaire; Diagnostic Test: Patient Health Questionnaire (PHQ-9); Diagnostic Test: Post Traumatic Stress Disorder questionnaire (PTSD-8); Diagnostic Test: Experiences in Close Relationship Scale questionnaire (ECR-S)

INTERVENTIONS:
Diagnostic Test: Generalized Anxiety Disorder-7 (GAD 7) — test that will evaluate persistent and excessive worry about a number of different things. People with Generalized Anxiety Disorder may anticipate disaster and may be overly concerned about money, health, family, work, or other issues. Individuals with Generalized Anxiety Disorder find it difficult to control their worry.
Diagnostic Test: Background questionnaire — questionnaire on the living conditions, socio-professional contexts and environmental conditions of the participants
Diagnostic Test: Impact of COVID-19 questionnaire — status of the patient with regard to the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2 virus)
Diagnostic Test: Confinement and Communication During the COVID-19 Pandemic — know the experience of containment and isolation during the pandemic
Diagnostic Test: Mental Health questionnaire — welfare effect
Diagnostic Test: Patient Health Questionnaire (PHQ-9) — assess depression during the pandemic
Diagnostic Test: Post Traumatic Stress Disorder questionnaire (PTSD-8) — Assessing the trauma of subjects during the pandemic
Diagnostic Test: Experiences in Close Relationship Scale questionnaire (ECR-S) — Measuring social ties and attachment of subjects

SUMMARY:
The aim of this project is to evaluate the impact of pandemic and nonconfinement related to anxiety and eventual immune diseases with several standardized questionnaires : Implant Stability Quotient (ISQ) , Generalized Anxiety Disorder-7 (GAD-7), Patient Health Questionnaire -9 (PHQ-9), Post Traumatic Stress Disorder-8 (PTSD-8), and Experiences in Close Relationship Scale (ECRS).

DETAILED DESCRIPTION:
The COVID-19 pandemic and prevention strategise have strongly impacted family lives, social lives, professional lives, and income; resulting in increased reporting of stress and anxiety within patients. This risk of infection 'post-confinement' is an additional source of stress for people returning to their professional and social lives. There are evidence showing a relationship between stress, immunity and the prognosis of several infections and inflammatory diseases.

The COVID-19 pandemic and prevention strategise have strongly impacted family lives and induced a high level of anxiety and other types of stress. This risk of infection 'post-confinement' is an additional source of stress for people returning to their professional and social life.

There are evidences showing a relationship between stress, immunity and the prognosis of several infections and inflammatory diseases.

The aim of this project is to launch an online survey that measures population stress felt during the pandemic and post-confinement time and possible effects on eventual immune mediated disorders (allergies, auto-immunity..) through the report of new events or flares. The stress will first be measured on standardized anxiety GAD-7scale but also on more parameters (ISQ, PHQ-9, PTSD-8, and ECR-S). Socio-economic and environmental parameters will be recorded.

Level of anxiety and other stress parameters as well as occurrence of inflammatory events will be measured according to the calendar and confinement /post confinement timing. Risk factors will be looked for, by multi parametric data analysis.

The survey has been built in a user-friendly, accessible way so the investigators can expect a high number of participants (at least 400), especially as people are highly concerned by the situation and will be motivated to take part.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteer who agreed to answer the questionnaires
* Age ≥ 18 years old
* Adult affiliated or having a duty to a social security scheme

Exclusion Criteria:

* Children under 18 years old
* Inability to understand information letter, consent, or to use online questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health Volunteers
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Results of the Generalized Anxiety Disorder (GAD-7) | 5 Minutes
  test that will evaluate persistent and excessive worry about a number of different things. People with Generalized Anxiety Disorder may anticipate disaster and may be overly concerned about money, health, family, work, or other issues. Individuals with Generalized Anxiety Disorder find it difficult to control their worry.
  Scored between 0-21:
  Cut offs:
  * 0-4 = None
  * 5-9 = Mild anxiety
  * 10-14 = Moderate anxiety
  * 15-21 = Severe anxiety

SECONDARY OUTCOMES:
Results of the Mental Health questionnaire | 5 minutes
  Welfare effect (mental health positively or negatively affected by COVID-19; why?) Scored between 7-42. These are treated as continuous variables.
Results of the Patient Health Questionnaire (PHQ-9) | 5 minutes
  assess depression during the pandemic
  Scored between 0-27:
  Cut offs:
  * 0-4 = None
  * 5-9 = Mild depression
  * 10-14 = Moderate depression
  * 15-19 = Moderately severe depression
  * 20-27 = Severe depression
Results of the Post Traumatic Stress Disorder (PTSD-8) | 5 minutes
  Assessing the trauma of subjects during the pandemic Scored between 7-42. These are treated as continuous variables.
Results of the Experiences in Close Relationship Scale questionnaire (ECR-S) | 5 minutes
  Measuring social ties and attachment of subjects Scored between 7-42. These are treated as continuous variables.

CONTACTS AND LOCATIONS:
Overall Officials: Claude LAMBERT, MD PhD HDR, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne, France
- Centre de Recherche et d'Innovation Clinique, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No